CLINICAL TRIAL: NCT02492282
Title: Evaluation of a Novel Closed-loop Propofol and Remifentanil System Guided by Bispectral Index Compared to a TCI Open-loop System: a Randomized Controlled Trial.
Brief Title: Evaluation of a Novel Closed-loop Propofol and Remifentanil System Guided by Bispectral Index Compared to a TCI Open-loop System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Fabian David Casas Arroyave, MD, Ms., Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIVA-15517889
Record Dates: First submitted 2015-07-04; First posted 2015-07-08 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia, General; Anesthesia, Intravenous
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed-Loop (Experimental): This group includes patients with randomization process be assigned to closed loop intravenous anesthesia; the system evaluates, feeds and acts according to the patient's bispectral index, excluding the anesthesiologist. This system use a variable control of specific therapeutic effect; a target value for this variable (set point); an actuator control (infusion pump), a system (patient) and a control algorithm.
  Interventions: Device: Closed-Loop propofol and remifentanil system by Bispectral Index; Drug: propofol
- Open-Loop (Active Comparator): This group includes patients with the randomization process are assigned to open loop in which the application of anesthetics is exclusively with pharmacokinetic parameters using TCI and employs mathematical models drug. For propofol used Schneider model and Minto model for remifentanil based on effective site concentration. Changes will be made by the anesthesiologist according to his criteria, trying to keep the BIS range of 40 and 60.
  Interventions: Device: Open-Loop propofol and remifentanil by Target Controlled Infusion; Drug: propofol

INTERVENTIONS:
Device: Closed-Loop propofol and remifentanil system by Bispectral Index
  Arms: Closed-Loop
Device: Open-Loop propofol and remifentanil by Target Controlled Infusion
  Arms: Open-Loop
Drug: propofol

SUMMARY:
Closed loop system in intravenous anesthesia is more effective to maintain depth of anesthesia compared with manual system open, it is unclear what driver and variables to achieve this goal be more physiological; in the literature doesn´t exist studies showing that the closed-loop system for both hypnotic and opioid is better than the controlled pharmacokinetic models and open loop system (target controlled infusion-TCI) to maintain anesthetic depth. In addition, the infusion of the opioid lacks physiological controllers in closed loop. Thus, a system was designed for intravenous anesthesia in closed loop for propofol as hypnotic based on neuromonitoring bispectral index as anesthetic depth, and was integrated an additional closed system for remifentanil using hemodynamic variables and control algorithm associated with bispectral index.

The purpose of this study is to determine the therapeutic effectiveness of a new system of administration of intravenous anesthesia in closed loop to maintain a depth of anesthesia compared to an open loop system TCI.

DETAILED DESCRIPTION:
Total intravenous anesthesia (TIVA) is a technique in which general anesthesia is administered intravenously, exclusively, a combination of drugs in the absence of any anesthetic agent inhaled1. TIVA development is closely linked to that of perfusion systems; these make total intravenous anesthesia enjoy several advantages as high hemodynamic stability, anesthetic depth more balanced, rapid and predictable recovery, less medication administered, less pollution and lower toxicity , not only for the patient also for the surgical equipment 2,3, 4 .

Two methods for controlling drug administration can be distinguished: open-loop and closed-loop control.

Open loop control applies pharmacokinetics (PK)/pharmacodynamics (PD) models based on the estimation of concentration of the drug in certain parts of the body, without measuring these concentrations in real time. The inaccuracy resulting from the absolute concentration requires the clinician to manually titrate dosage and objective observation based on the concentration of the desired therapeutic effect. This titration requires high clinical experience and a process of intensive monitoring, which may divert the attention from critical situations which in turn leads to suboptimal therapy or even to put safety at risk patient5, 6.

The application of closed-loop systems for the administration of an anesthetic requires a perfect balance of all the basic components of a system of this type: a variable control of the specific therapeutic effect; a target value for this variable (usually called set point); an actuator control (in this case, the drug infusion pump); a system (in this case the patient); and control algorithm7. This system excludes the control anesthesiologist drug infusion which is determined by one or more clinical variables that directly reflect the relationship PK / PD which previously established the attending anesthesiologist. The controller automatically calculates the optimal rate of infusion based on the current value and the desired value of the controlling variable and previously established mathematical models.

With the appearance of electroencephalographic monitoring practice as a control variable, began to conduct studies to assess the cerebral effect of anesthetics. Linear model two compartments is used to describe the relationship of drug concentration and an adaptive controller and this system was used subsequently using EEG to study the interaction of opioid and propofol 8,9. After marketing bispectral index derived from the EEG, began to evaluate closed loop systems using the BIS technology in several studies concluding that such systems not only makes more predictable anesthetic depth, but provides greater intraoperative hemodynamic stability and early recovery of the sedative and hypnotic effects of propofol 10,11,12,13,14.

Closed loop system in intravenous anesthesia is more effective to maintain the depth of anesthesia compared with manual system open, it is unclear what the driver and the variables to achieve this goal be more physiological and accurately; in the literature doesn´t exist studies showing that the closed-loop system for both hypnotic and opioid is better than the controlled pharmacokinetic models and open loop system to maintain anesthetic depth. In addition, the infusion of the opioid lacks physiological controllers in closed loop. Thus, a system was designed for intravenous anesthesia in closed loop for propofol as hypnotic based on neuromonitoring bispectral index as anesthetic depth, and was integrated an additional closed system for remifentanil using hemodynamic variables and control algorithm associated with bispectral index.

The purpose of this study is to determine the therapeutic effectiveness of a new system of administration of intravenous anesthesia in closed loop to maintain a depth of anesthesia compared to an open loop system TCI.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Scheduled for noncardiac surgery elective low-risk or intermediate
* Expected surgery time greater than 1 hour
* Procedure requiring general anesthesia
* Classification of the American Society of Anesthesiologists (ASA) as I or II

Exclusion Criteria:

* Pregnant women
* Surgery scheduled urgent or emergency
* Personal history of allergy to eggs or any other part of propofol
* Personal history of abnormalities or congenital or acquired cognitive sequels: infantile cerebral palsy, Down syndrome, cerebral ischemic disease, traumatic brain injury, brain tumor, autism.
* Chronic use of benzodiazepines or antipsychotics
* A patient who does not consent to participate in the study prior to surgery or before randomization
* Need for anesthetic or analgesic blockade before surgery peripheral nerve

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Time in adequate anesthetic depth | intraoperative
  Difference in therapeutic effectiveness determined by the time in state suitable anesthetic depth. The proper anesthetic depth is defined as the efficacy to maintain a Bispectral Index in the range of 40 - 60 during a surgery.

SECONDARY OUTCOMES:
Proportion of patients with adequate anesthetic depth | intraoperative
  Difference in the proportion of patients with adequate depth of anesthesia. Anesthetic depth is defined as appropriate when the percentage of time the patient spends in this range (BIS between 40 and 60) is greater than 80%.
Difference in technical performance drivers intravenous infusion | intraoperative
  The performance will be determined using methods Varvel et al. Performance error (PE) is defined as the difference between the actual value and the target value. Median performance error (MDPE) and Error Performance Absolute Median (MDAPE) as measures of validity and accuracy, respectively. Wobble as a measure of variability in performance error.
Difference in the proportion of patients with adequate intraoperative analgesia | intraoperative
  Difference in the proportion of patients with adequate analgesia intraoperative defined according to the values of "analgoscore", a scale for the measurement of intraoperative pain developed and validated by Hemmerling et al. It is based on measuring the averagely nociception determined mean arterial pressure and heart rate, which generates a numerical range between -9 and 9. A value between -3 and +3 represents excellent pain control; a value between -6 to -3 and +3 to +6 indicates good pain control;-6 To -9 and +9 +6 it indicates inadequate pain control. Adequate intraoperative analgesia is considered when the percentage of time the patient spends in the range of values between - 6 and +6 is greater than 80%.
Difference in the proportion of patients in which they have to perform manual modification of the drug infusion. | intraoperative
  Any manual handling of the anesthesia system is considered one that performs different from the initial programming output.
Difference in the rate of change of an intravenous anesthetic technique to a technique based on halogenated. | intraoperative
Amount of anesthetic medications used during the anesthetic | intraoperative
Proportion of patients with haemodynamic instability. | intraoperative
  Hemodynamic instability any of the following events are considered: Reduction of more than 20% of the basal MAP and HR increased more than 10% of baseline; Decreased heart rate less than 10% increase in MAP and more than 5%; Need for vasopressor support with bolus or continuous infusion of drugs alpha and / or beta-agonists; Parasympatholytic need.
Proportion of patients with intraoperative recall | 2 hours after surgery
  Difference in the proportion of patients with intraoperative recall. Intraoperative recall will be measured with a validated scale as Michigan scale, which ranks intraoperative recall in 6 classes: Class 0, where there are no symptoms of memory; Class 1, isolated auditory perceptions; Class 2, tactile perceptions, such as surgical manipulation or endotracheal intubation; Class 3, Pain; Class 4, paralysis defined as the feeling of being unable to move, speak or breathe; Class 5, paralysis and pain. If any of these classes is associated with negative emotional impact (fear, anxiety, suffocation feeling of death, etc.) will be added to the letter D
Proportion of patients with awakening during anesthetic maintenance | intraoperative
  It will be as any episode of patient movement during surgical painful stimulus including upper, lower or respiratory system (cough reflex to the presence of the endotracheal tube) extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Casas, MD, Ms, Principal Investigator — Universidad de Antioquia
Locations (1):
- Hospital Universitario San Vicente Fundación, Medellín, Antioquia, Colombia

REFERENCES:
- [Background] Carregal A, Lorenzo A, Taboada JA, Barreiro JL. [Intraoperative control of mean arterial pressure and heart rate with alfentanyl with fuzzy logic]. Rev Esp Anestesiol Reanim. 2000 Mar;47(3):108-13. Spanish. PMID 10800361
- [Result] Ngan Kee WD, Khaw KS, Ng FF, Tam YH. Randomized comparison of closed-loop feedback computer-controlled with manual-controlled infusion of phenylephrine for maintaining arterial pressure during spinal anaesthesia for caesarean delivery. Br J Anaesth. 2013 Jan;110(1):59-65. doi: 10.1093/bja/aes339. Epub 2012 Sep 25. PMID 23015618
- [Result] Janda M, Simanski O, Bajorat J, Pohl B, Noeldge-Schomburg GF, Hofmockel R. Clinical evaluation of a simultaneous closed-loop anaesthesia control system for depth of anaesthesia and neuromuscular blockade*. Anaesthesia. 2011 Dec;66(12):1112-20. doi: 10.1111/j.1365-2044.2011.06875.x. Epub 2011 Sep 23. PMID 21950720
- [Result] Liu N, Chazot T, Trillat B, Pirracchio R, Law-Koune JD, Barvais L, Fischler M. Feasibility of closed-loop titration of propofol guided by the Bispectral Index for general anaesthesia induction: a prospective randomized study. Eur J Anaesthesiol. 2006 Jun;23(6):465-9. doi: 10.1017/S0265021506000196. PMID 16672092
- [Result] Sakai T, Matsuki A, White PF, Giesecke AH. Use of an EEG-bispectral closed-loop delivery system for administering propofol. Acta Anaesthesiol Scand. 2000 Sep;44(8):1007-10. doi: 10.1034/j.1399-6576.2000.440819.x. PMID 10981581
- [Result] De Smet T, Struys MM, Neckebroek MM, Van den Hauwe K, Bonte S, Mortier EP. The accuracy and clinical feasibility of a new bayesian-based closed-loop control system for propofol administration using the bispectral index as a controlled variable. Anesth Analg. 2008 Oct;107(4):1200-10. doi: 10.1213/ane.0b013e31817bd1a6. PMID 18806028
- [Result] Puri GD, Kumar B, Aveek J. Closed-loop anaesthesia delivery system (CLADS) using bispectral index: a performance assessment study. Anaesth Intensive Care. 2007 Jun;35(3):357-62. doi: 10.1177/0310057X0703500306. PMID 17591128
- [Result] Struys MM, De Smet T, Versichelen LF, Van De Velde S, Van den Broecke R, Mortier EP. Comparison of closed-loop controlled administration of propofol using Bispectral Index as the controlled variable versus "standard practice" controlled administration. Anesthesiology. 2001 Jul;95(1):6-17. doi: 10.1097/00000542-200107000-00007. PMID 11465585
- [Result] Hemmerling TM, Arbeid E, Wehbe M, Cyr S, Taddei R, Zaouter C. Evaluation of a novel closed-loop total intravenous anaesthesia drug delivery system: a randomized controlled trial. Br J Anaesth. 2013 Jun;110(6):1031-9. doi: 10.1093/bja/aet001. Epub 2013 Feb 20. PMID 23427212